CLINICAL TRIAL: NCT01373099
Title: Articulating Versus Static Antibiotic Loaded Spacers for the Treatment of Prosthetic Hip Infection
Brief Title: Study of Antibiotic Spacer Design to Treat Infection After Hip Replacement
Acronym: SPACERHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Thomas Jefferson University (Other); Central DuPage Hospital (Other)
Responsible Party: Principal Investigator, Peter N. Chalmers, MD, Resident, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACERHIP
Record Dates: First submitted 2011-06-06; First posted 2011-06-14 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis; Hip Infection; Prosthetic Joint Infection; Complications; Arthroplasty, Infection or Inflammation; Complications; Arthroplasty
Keywords: arthroplasty; hip replacement; Osteoarthritis; knee Infection; Prosthetic Joint Infection; Complications; Arthroplasty, Infection or Inflammation; Complications; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static Spacer (Experimental): Patients in this group will be randomized to a static, nonarticulating, antibiotic-impregnated cement spacer.
  Interventions: Procedure: Implantation of a static, non-articulating cement spacer.
- Articulating spacer (Experimental): Patients in this group will be randomized to an articulating antibiotic-impregnated cement spacer.
  Interventions: Procedure: Implantation of an articulating spacer.

INTERVENTIONS:
Procedure: Implantation of a static, non-articulating cement spacer. — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed using 3.0 g of Vancomycin and 1.0 g of Tobramycin for each 40 g packet of cement. Static spacers will be hand-made with a rod of antibiotic-impregnated cement and cement beads of sufficient quantity to fill the acetabulum.
  Arms: Static Spacer
Procedure: Implantation of an articulating spacer. — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed using 3.0 g of Vancomycin and 1.0 g of Tobramycin for each 40 g packet of cement. Articulating spacers will be formed of antibiotic-impregnated cement using the Stage One system (Biomet, Warsaw, IN) sized to fit the endosteal and acetabular bone defect.
  Arms: Articulating spacer

SUMMARY:
Infection remains one of the most difficult-to-treat complications of total hip arthroplasty. The gold standard treatment is two-stage removal of the prosthesis with later replacement of permanent implants.The first stage consists of removal of the infected arthroplasty components and the surrounding devitalized tissue, copious pulsed irrigation, and placement of a temporary antibiotic-impregnated cement spacer. This spacer is typically left in place six weeks, during which time the patient receives intravenous antibiotics. After the surgeon feels that the infection has been eradicated, or if a second debridement is required, a second operative procedure is performed. While the use of an antibiotic spacer is well accepted, whether the spacer should immobilize the hip (a so-called "static" spacer) or allow for range of motion (a so-called "articulating" spacer) is controversial. Proponents of static spacers argue that immobilization of the periarticular soft tissues aids in clearance of the infection and that these spacers are simpler to fashion intraoperatively. Proponents of articulating spacers argue that they improve hip function, prevent damage to the musculature surrounding the hip, allow easier reimplantation, improve hip function, and prevent dislocation following hip reimplantation. While good results have been described with both methods, comparative trials have been conflicting as to whether spacer design alters hip function, operative time, and dislocation rates. Equipoise exists within the literature, and no randomized clinical trial has been conducted to evaluate this issue.

The purpose of this study is to compare articulating and static antibiotic-impregnated spacers for the treatment of chronic periprosthetic infection complicating total hip arthroplasty through a prospective, randomized clinical trial. The goals of this trial are to determine the effect of spacer design upon eradication of infection, hip function, ease of reimplantation, and dislocation rates. The investigators hypothesize that articulating spacers will provide shorter operative times at replantation while improving hip function and hip dislocation rates following hip reimplantation.

DETAILED DESCRIPTION:
After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed using 3.0 g of Vancomycin and 1.0 g of Tobramycin for each 40 g packet of cement. Articulating spacers will be formed of antibiotic-impregnated cement using the Stage One system (Biomet, Warsaw, IN) sized to fit the endosteal and acetabular bone defect. Static spacers will be hand-made with a rod of antibiotic-impregnated cement and cement beads of sufficient quantity to fill the acetabulum.

Post-operatively, all patients will be made touch-down weight bearing protected with a walker or crutches. At the time of reimplantation, the joint will be aspirated and multiple cultures obtained along with intraoperative histopathological analysis to evaluate for persistent infection.

Data collected preoperatively will include age, gender, laterality, etiology of hip degeneration, comorbidities, Harris Hip score, infecting organisms and Paprosky femoral and acetabular bone loss classification. The Harris Hip score has been used extensively in the study of revision hip arthroplasty and has been found to be reliable and valid and will be determined preoperatively and at all follow-up visits.

Data collected at the time of implant removal and reimplantation will include operative time, blood loss, surgical approach, and need for an extended trochanteric osteotomy. Radiographs performed immediately following and just prior to reimplantation will be reviewed to determine if the spacer utilized has caused bone loss; bone loss to the cut bony surfaces will be confirmed intraoperatively. At each follow-up visits radiographic appearance, the Harris Hip Score, dislocation events, recurrence of infection, and the need for revision or reoperation of any kind on the hip will be determined.

All portions of this study will be part of conventional care except for randomization and collection of the Harris Hip Score. Which type of spacer is used currently depends upon the judgment of the attending surgeons and both are used routinely.

The primary outcome variable will be Harris Hip Score. A power analysis was conducted with the assistance of Dr. Mario Moric at Rush. Using the standard deviation of Harris Hip Scores from Hsieh and colleagues (2004) and Fehring and colleagues (1999), the largest previous studies reporting such data, Dr. Moric estimated 56 patients, 28 patients per group, would be needed to detect a clinically relevant difference of ten points. To account for attrition, our target total sample size will be 80 patients.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosis of periprosthetic joint infection of a primary total hip arthroplasty with a planned two-stage exchange procedure.

Exclusion Criteria:

1. Infection of a revision as opposed to a primary total hip arthroplasty
2. Medically unfit for operative intervention
3. Extensive bone loss preventing the use of an articulating spacer
4. Soft-tissue defects that prevent the use of an articulating spacer
5. Known allergy to polymethylmethacrylate, tobramycin or vancomycin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | outcome will be collected until 2 years post-operatively
  The Harris Hip score has been used extensively in the study of revision hip arthroplasty and has been found to be reliable and valid to determine hip arthroplasty outcomes.

SECONDARY OUTCOMES:
Operative time | at the time of spacer revision, which would be up to a maximumup to 2 years after patient enrollment
Hip dislocation rates | outcomes will be collected until 2 years post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center; Scott Sporer, MD, Principal Investigator — Rush University Medical Center; Peter Chalmers, MD, Principal Investigator — Rush University Medical Center; Javad Parvizi, MD, Principal Investigator — Thomas Jefferson Hospital; Matt Austin, MD, Principal Investigator — Thomas Jefferson Hospital
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Kurtz SM, Lau E, Schmier J, Ong KL, Zhao K, Parvizi J. Infection burden for hip and knee arthroplasty in the United States. J Arthroplasty. 2008 Oct;23(7):984-91. doi: 10.1016/j.arth.2007.10.017. Epub 2008 Apr 10. PMID 18534466
- [Background] Peersman G, Laskin R, Davis J, Peterson M. Infection in total knee replacement: a retrospective review of 6489 total knee replacements. Clin Orthop Relat Res. 2001 Nov;(392):15-23. PMID 11716377
- [Background] Della Valle CJ, Paprosky WG. The femur in revision total hip arthroplasty evaluation and classification. Clin Orthop Relat Res. 2004 Mar;(420):55-62. doi: 10.1097/00003086-200403000-00009. PMID 15057079
- [Background] Biring GS, Kostamo T, Garbuz DS, Masri BA, Duncan CP. Two-stage revision arthroplasty of the hip for infection using an interim articulated Prostalac hip spacer: a 10- to 15-year follow-up study. J Bone Joint Surg Br. 2009 Nov;91(11):1431-7. doi: 10.1302/0301-620X.91B11.22026. PMID 19880885
- [Background] Hsieh PH, Shih CH, Chang YH, Lee MS, Shih HN, Yang WE. Two-stage revision hip arthroplasty for infection: comparison between the interim use of antibiotic-loaded cement beads and a spacer prosthesis. J Bone Joint Surg Am. 2004 Sep;86(9):1989-97. PMID 15342762
- [Background] Younger AS, Duncan CP, Masri BA, McGraw RW. The outcome of two-stage arthroplasty using a custom-made interval spacer to treat the infected hip. J Arthroplasty. 1997 Sep;12(6):615-23. doi: 10.1016/s0883-5403(97)90133-9. PMID 9306211
- [Background] Anagnostakos K, Wilmes P, Schmitt E, Kelm J. Elution of gentamicin and vancomycin from polymethylmethacrylate beads and hip spacers in vivo. Acta Orthop. 2009 Apr;80(2):193-7. doi: 10.3109/17453670902884700. PMID 19404802
- [Background] Fink B, Rechtenbach A, Buchner H, Vogt S, Hahn M. Articulating spacers used in two-stage revision of infected hip and knee prostheses abrade with time. Clin Orthop Relat Res. 2011 Apr;469(4):1095-102. doi: 10.1007/s11999-010-1479-1. Epub 2010 Jul 28. PMID 20665141
- [Background] Lewis G. Alternative acrylic bone cement formulations for cemented arthroplasties: present status, key issues, and future prospects. J Biomed Mater Res B Appl Biomater. 2008 Feb;84(2):301-19. doi: 10.1002/jbm.b.30873. PMID 17588247
- [Background] Affatato S, Mattarozzi A, Taddei P, Robotti P, Soffiatti R, Sudanese A, Toni A. Investigations on the wear behaviour of the temporary PMMA-based hip Spacer-G. Proc Inst Mech Eng H. 2003;217(1):1-8. doi: 10.1243/095441103762597665. PMID 12578213
- [Background] Gooding CR, Masri BA, Duncan CP, Greidanus NV, Garbuz DS. Durable infection control and function with the PROSTALAC spacer in two-stage revision for infected knee arthroplasty. Clin Orthop Relat Res. 2011 Apr;469(4):985-93. doi: 10.1007/s11999-010-1579-y. PMID 20878287
- [Background] Haddad FS, Masri BA, Campbell D, McGraw RW, Beauchamp CP, Duncan CP. The PROSTALAC functional spacer in two-stage revision for infected knee replacements. Prosthesis of antibiotic-loaded acrylic cement. J Bone Joint Surg Br. 2000 Aug;82(6):807-12. doi: 10.1302/0301-620x.82b6.10486. PMID 10990301
- [Background] Wentworth SJ, Masri BA, Duncan CP, Southworth CB. Hip prosthesis of antibiotic-loaded acrylic cement for the treatment of infections following total hip arthroplasty. J Bone Joint Surg Am. 2002;84-A Suppl 2:123-8. doi: 10.2106/00004623-200200002-00017. No abstract available. PMID 12479350
- [Background] Fehring TK, Odum S, Calton TF, Mason JB. Articulating versus static spacers in revision total knee arthroplasty for sepsis. The Ranawat Award. Clin Orthop Relat Res. 2000 Nov;(380):9-16. doi: 10.1097/00003086-200011000-00003. PMID 11064968
- [Background] Paprosky WG, Perona PG, Lawrence JM. Acetabular defect classification and surgical reconstruction in revision arthroplasty. A 6-year follow-up evaluation. J Arthroplasty. 1994 Feb;9(1):33-44. doi: 10.1016/0883-5403(94)90135-x. PMID 8163974
- [Background] Shields RK, Enloe LJ, Evans RE, Smith KB, Steckel SD. Reliability, validity, and responsiveness of functional tests in patients with total joint replacement. Phys Ther. 1995 Mar;75(3):169-76; discussion 176-9. doi: 10.1093/ptj/75.3.169. PMID 7870749
- [Background] Soderman P, Malchau H. Is the Harris hip score system useful to study the outcome of total hip replacement? Clin Orthop Relat Res. 2001 Mar;(384):189-97. doi: 10.1097/00003086-200103000-00022. PMID 11249165
- [Background] Fehring TK, Calton TF, Griffin WL. Cementless fixation in 2-stage reimplantation for periprosthetic sepsis. J Arthroplasty. 1999 Feb;14(2):175-81. doi: 10.1016/s0883-5403(99)90122-5. PMID 10065723
- [Derived] Nahhas CR, Chalmers PN, Parvizi J, Sporer SM, Deirmengian GK, Chen AF, Culvern CN, Moric M, Della Valle CJ. Randomized Trial of Static and Articulating Spacers for Treatment of the Infected Total Hip Arthroplasty. J Arthroplasty. 2021 Jun;36(6):2171-2177. doi: 10.1016/j.arth.2021.01.031. Epub 2021 Jan 21. PMID 33581975